CLINICAL TRIAL: NCT05598125
Title: Comparative Investigation of the One-time Use of an Electronic Cigarette (E-cigarette) Versus a Normal Tobacco Cigarette on Vascular Function in Healthy Male Smokers
Brief Title: Study of Vascular Function Before vs After Smoking an E-cigarette as Compared to a Normal Cigarette
Acronym: ECIG-8
Status: Terminated | Type: Observational
Why Stopped: due to recruitment reasons the study was prematurely ended
Sponsor: GWT-TUD GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: ECIG-8
Record Dates: First submitted 2019-08-01; First posted 2022-10-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2019-08

CONDITIONS: Endothelial Function
Keywords: arterial wave reflection; microvascular function; e-cigarette
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Brachial artery diameter change in response to reactive hyperemia (flow-mediated vasodilation, %)
  * Circulating biomarkers of endothelial function and damage (endothelin-1; BH4/BH2)
  * Augmentation index in response to salbutamol and glyceryl trinitrate (%),
  * Retinal arterial and venous diameter in response to flicker-light stimulation (%)
  * Central retinal arterial and venous equivalent (CRAE, CRVE) and arteriolar-to-venular ratio (AVR)
  * Functional in vitro assays and gene expression studies (endothelial nitric oxide synthase (eNOS), NRF2 pathway and target genes (HMOX1, NQO1); adhesion molecules (ICAM1, VCAM1, SELE, CCL2))
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Smoker_1: Begins with e-cigarette crosses over to conventional cigarette
  Interventions: Device: electronic cigarette (e-cigarette); Device: conventional tobacco cigarette
- Non smoker: never smoking participants as control group
- Smoker_2: Begins with conventional cigarette crosses over to e-cigarette
  Interventions: Device: electronic cigarette (e-cigarette); Device: conventional tobacco cigarette

INTERVENTIONS:
Device: electronic cigarette (e-cigarette)
  Groups: Smoker_1; Smoker_2
Device: conventional tobacco cigarette
  Groups: Smoker_1; Smoker_2

SUMMARY:
Investigation of the effect of one-time use of an electronic e-cigarette in comparison to smoking a conventional cigarette on in vivo conduit endothelial function in healthy long-term smokers

DETAILED DESCRIPTION:
The overall aim of this study is to compare the short-term vascular effects of smoking an e-cigarette versus smoking a conventional tobacco cigarette in vivo and in vitro.

The specific objectives are as follows:

i. To evaluate the effects of e-cigarette and conventional combustible cigarette (CCC) use on microvascular and macrovascular endothelial function and stiffness in healthy smokers.

ii. To assess circulating markers of endothelial function in response to e-cigarette and CCC smoking.

iii. To investigate the vascular effects of e-cigarette and CCC use on a molecular level by exposing endothelial cells with stimulated serum from the intervention study.

Primary Objective and Outcome Parameter:

The primary objective of this investigator initiated trial (IIT) is to evaluate the short-term effect of e-cigarette puffing on conduit artery function in comparison to smoking a CCC in healthy male long-term smokers.

The relative change in brachial artery diameter in response to reactive hyperemia (flow-mediated vasodilation), a validated surrogate marker of conduit endothelial function, will be used as primary endpoint. FMD [%] is defined as (brachial diameter 60 s after cuff deflation [mm] - baseline brachial diameter [mm]) x 100 / baseline brachial diameter [mm].

The primary outcome measure is the absolute difference of FMD after e-cigarette and CCC.

Secondary Objective and Outcome Parameter:

The secondary objectives are to evaluate in vivo endothelial function in other vascular beds, especially in the microcirculation and the systemic circulation, as well as other aspects of vascular function like stiffness of the arterial tree. Endothelial dysfunction, a key event of atherosclerosis development, is characterized by a respective increase or decrease of endothelium-derived molecules and changes in upstream signaling pathways that control the synthesis and bioavailability of these endothelium-derived molecules. Analysis of circulating biomarkers of endothelial function and expression studies of enzymes involved in endothelial activation will help to closely characterize possible effects of e-cigarette exposure on in vivo endothelial function.

Secondary endpoints are:

* Augmentation index in response to salbutamol (%) as surrogate of global endothelial function in relation to its response to glyceryl trinitrate (%)
* Augmentation index (%) as marker of pulse wave reflection and stiffness
* Retinal arterial and venous diameter in response to flicker-light stimulation (%) as surrogate of microvascular endothelial function
* Central retinal arterial and venous equivalent and arteriolar-to-venular ratio as indicators of generalized arterial narrowing
* Circulating biomarkers of endothelial function and activation (Endothelin-1; BH4/BH2) Secondary outcome measures are the absolute differences of secondary endpoints between e-cigarette and CCC (refer to section 13.4.2).

Functional in vitro assays and molecular analyses:

* mRNA and protein expression of endothelial nitric oxide synthase (eNOS), NRF2 target genes HMOX1, NQO1 and adhesion molecules (ICAM1, VCAM1, SELE, CCL2).
* Primary cultures of human umbilical vein endothelial cells will be stimulated with serum of human subjects (sampled before or after smoking of one cigarette or e-cigarette) and potential of wound healing will be determined.

Tertiary Objective and Outcome Parameter:

The tertiary objective is to assess differences in vascular function between smokers and never smokers. Tertiary endpoints are baseline values of primary and secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* • Subjects must be males between 22 and 35 years of age, inclusive.

  * Subjects must be able to comprehend, sign and date a written informed consent prior to entering the study.
  * Subjects must be willing and able to comply with the protocol requirements for the duration of the study.
  * Subjects must have experienced one of the following:

    * Smoked for at least the last 4 years and at least 5 cigarettes a day or 1 pack-years,
    * Never having regularly smoked, i.e. < 20 cigarettes in their lifetime and not in last 5 years.

Exclusion Criteria:

* Consumption of cigars, other tobacco and nicotine products and light-cigarettes (less than 8 mg ISO tar).

  * Exhaled CO levels < 10 ppm (smokers) and ≥ 10 ppm (never smokers).
  * Urinary cotinine < 200 ng/ml for smoker group
  * Treatment for arterial hypertension, or clinic blood pressure ≥140/90 mmHg.
  * Body mass index ≥ 30 kg/m2
  * Ocular diseases, glaucoma.
  * Convulsive disorder/epilepsy or intake of anticonvulsant drugs.
  * Subjects with a clinically significant or unstable medical or surgical condition that would preclude safe and complete study participation, as determined by medical history, physical exams, ECG, abnormal laboratory tests. Such conditions may include hepatic, renal or metabolic diseases, systemic disease, acute infection, current malignancy or recent history (5 years) of malignancy, major psychiatric disorder, history of drug and/or alcohol abuse and allergies that could be detrimental according to the investigator's judgment.
  * Prior participation in a clinical study in last 4 weeks.
  * Intake of drugs with potential impact on the endothelial function resp. autonomic nervous system.
  * Known intolerance against salbutamol, nitroglycerin and/or propylene glycol.
  * Regular intake of vitamins and mineral supplements.
  * Heavy exercisers and trained athletes (> 5 hours physical activity / week).

Ages: 22 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 80 smokers 25 never smokers will be additionally recruited as a control group who will undergo the same measurements and analyses without smoking intervention.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
change in conduit artery function related to the smoking pattern | 7 days
  Conduit artery function is defined as the relative response of brachial artery diameter to reactive hyperemia termed as flow-mediated vasodilation (FMD). The primary outcome measure is the absolute difference of FMD after e-cigarette and conventional cigarette consume

SECONDARY OUTCOMES:
Retinal arterial and venous diameter in response to flicker-light stimulation (%) as surrogate of microvascular endothelial function | 7 days
  Secondary outcome measures are the absolute differences of secondary endpoints between e-cigarette and CCC
Change in CRAE (central retinal arteriolar equivalents) | 7 days
  To assess circulating marker of endothelial function in response to e-cigarette and CCC smoking.
  Central retinal arteriolar as marker of retinal structural microvascular abnormalities esp. generalized arteriolar narrowing and venular widening CRAE [µm]: will be automatically determined
Change in CRVE (central retinal venular equivalents) | 7 days
  To assess circulating marker of endothelial function in response to e-cigarette and CCC smoking.
  Central retinal venular equivalents as marker of retinal structural microvascular abnormalities esp. generalized arteriolar narrowing and venular widening CRVE [µm]: will be automatically determined
Change in AVR (arteriolar-to-venular ratio) | 7 days
  To assess circulating marker of endothelial function in response to e-cigarette and CCC smoking.
  Arteriolar-to-venular ratio as marker of retinal structural microvascular abnormalities esp. generalized arteriolar narrowing and venular widening AVR: will be automatically determined
Change in circulating biomarkers of endothelial function and activation - Endothelin-1 | 7 days
  To assess circulating marker of endothelial function in response to e-cigarette and CCC smoking.
  Endothelin-1 [pg/ml]
Change in circulating biomarkers of endothelial function and activation - BH4/BH2 | 7 days
  To assess circulating marker of endothelial function in response to e-cigarette and CCC smoking.
  BH4/BH2
Augmentation index in response to salbutamol (%) as surrogate of global endothelial function in relation to its response to glyceryl trinitrate (%) | 7 days
  Secondary outcome measures are the absolute differences of secondary endpoints between e-cigarette and CCC
Augmentation index (%) as marker of pulse wave reflection and stiffness | 7 days
  Secondary outcome measures are the absolute differences of secondary endpoints between e-cigarette and CCC

CONTACTS AND LOCATIONS:
Overall Officials: Tjalf Ziemssen, PhD, MD, Study Director — Zentrum für Klinische Neurowissenschaften, TU-Dresden; Henning Morawietz, PhD, Study Director — Bereich Gefäßendothel/Mikrozirkulation, TU-Dresden